CLINICAL TRIAL: NCT02644343
Title: Safety and Efficacy of Remote Programming of Nucleus Cochlear Implants
Acronym: TEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM 5650
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Remote Programming Group (Experimental): Subjects will undergo remote programming of Nucleus cochlear implants via Custom Sound software using an online interactive meeting platform.
  The intervention is the programming of the cochlear implant, the experimental aspect is the remote delivery method.
  Interventions: Device: Custom Sound

INTERVENTIONS:
Device: Custom Sound — Custom Sound is the programming software used to program Nucleus cochlear implants.

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of Nucleus cochlear implant programming via telecommunication.

DETAILED DESCRIPTION:
Cochlear implant recipients will undergo remapping at a location remote from their audiologist via telehealth. Audiologists will use an internet meeting platform to remotely log into the subject's computer and control the programming software. Remote programming sessions will be completed both with and without the assistance of a trained facilitator, and speech understanding will be tested in between mapping sessions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged greater than 12 years that are native English speakers and are capable of completing the study evaluation as deemed by their primary audiologist
* Unilateral or bilateral cochlear implant recipients of a CI24RE, CI422 or CI500 series implant who are in possession of a backup sound processor
* A minimum of 12 months' experience with a CP800 or CP900 series sound processor, and current MAP programmed within 12 months prior to Visit 1
* Willingness to participate in and to comply with all requirements of the protocol
* Able to demonstrate protocol competence as confirmed by primary audiologist

Exclusion Criteria:

* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations of remote service delivery
* Unwillingness or inability of the candidate to comply with all investigational requirements
* Additional handicaps that would prevent or restrict participation in the audiological evaluations
* Inability to demonstrate basic technological skills for simple computer-based tasks and device connecting after training by primary audiologist

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- [Background] PETERSON GE, LEHISTE I. Revised CNC lists for auditory tests. J Speech Hear Disord. 1962 Feb;27:62-70. doi: 10.1044/jshd.2701.62. No abstract available. PMID 14485785
- [Background] Wesarg T, Wasowski A, Skarzynski H, Ramos A, Falcon Gonzalez JC, Kyriafinis G, Junge F, Novakovich A, Mauch H, Laszig R. Remote fitting in Nucleus cochlear implant recipients. Acta Otolaryngol. 2010 Dec;130(12):1379-88. doi: 10.3109/00016489.2010.492480. Epub 2010 Jun 30. PMID 20586675
- [Background] McElveen JT Jr, Blackburn EL, Green JD Jr, McLear PW, Thimsen DJ, Wilson BS. Remote programming of cochlear implants: a telecommunications model. Otol Neurotol. 2010 Sep;31(7):1035-40. doi: 10.1097/MAO.0b013e3181d35d87. PMID 20147864

RESULTS

PARTICIPANT FLOW:
Groups:
- Remote Programming Group: Subjects will undergo remote programming of Nucleus cochlear implants via Custom Sound software using an online interactive meeting platform.
  The intervention is the programming of the cochlear implant, the experimental aspect is the remote delivery method.
  Custom Sound: Custom Sound is the programming software used to program Nucleus cochlear implants.
Period: Overall Study
Arm/Group | Remote Programming Group
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Remote Programming Group
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
Internal Implant Model [Count of Participants; unit: Participants]
  CI24R | 3
  CI24RE | 23
  CI422 | 8
  CI500 series | 6
Sound Processor Model [Count of Participants; unit: Participants]
  Nucleus 5 | 17
  Nucleus 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Speech Perception on Monosyllabic Word Test, CNC Words
Description: Subjects will listen to and repeat monosyllabic words from the Consonant Nucleus Consonant word test measured by percentage of words correct to examine their speech perception abilities after each remote programming session.
Time Frame: 2-4 weeks post remote programming session
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Remote Programming Group
Number analyzed (Participants) | 39
percentage of words correct
  Live Audiologist MAP | 70.5 (18.6)
  Facilitated Remote MAP | 72.4 (18.7)
  Unassisted Remote MAP | 72.5 (21.3)

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Remote Programming Group
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Programming Group (N=40)
Car Accident (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT02644343/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT02644343/SAP_001.pdf